CLINICAL TRIAL: NCT03859700
Title: EPITOPE Open-label Extension Study to Evaluate the Long-term Clinical Benefit and Safety of DBV712 in Peanut-Allergic Children
Brief Title: Follow-up of the EPITOPE Study to Evaluate Long-term Efficacy and Safety of DBV712 in Young Children
Acronym: EPOPEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOPEX (V712-305)
Record Dates: First submitted 2019-02-19; First posted 2019-03-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Peanut Allergy
Keywords: EPIT; Epicutaneous; Immunotherapy; Viaskin
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DBV712 250mcg (Experimental)
  Interventions: Biological: DBV712 250 mcg

INTERVENTIONS:
Biological: DBV712 250 mcg — DBV712 250 mcg, once daily

SUMMARY:
Open-label, follow-up study for subjects who completed the EPITOPE study.

ELIGIBILITY:
Inclusion Criteria:

* completion of the EPITOPE study

Exclusion Criteria:

* Generalized dermatologic disease (for example, active atopic dermatitis, uncontrolled generalized active eczema, ichthyosis vulgaris) extending widely on the skin and especially on the back or arms with no intact zones to apply the Viaskin patches.
* Diagnosis of asthma that evolved to severe, unstable or uncontrolled asthma

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects reaching an ED ≥1000 mg | 12 months
Proportion of subjects reaching an ED ≥1000 mg | 24 months
Proportion of subjects reaching an ED ≥1000 mg | 36 months

SECONDARY OUTCOMES:
Adverse Events (AEs), Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) | Throughout the study during 36 months

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Banner University Medical Center Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - David Geffen School of Medicine at University of California Los Angeles, Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Health Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Comer Children's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Childrens' Hospital, Boston, Massachusetts
  - University of Michigan - Allergy Specialty Clinic and Food Allergy Clinic, Ann Arbor, Michigan
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - The University of North Carolina - Chapell Hill, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Allergy & Asthma Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greenhawt M, Albright D, Anvari S, Arends N, Arkwright PD, Begin P, Blumchen K, Brown-Whitehorn T, Cassell H, Chan ES, Ciaccio CE, Deschildre A, Divaret-Chauveau A, Dorris S, Dorsey M, Du Toit G, Eiwegger T, Erlewyn-Lajeunesse M, Fleischer DM, Ford LS, Garcia-Lloret M, O'B Hourihane J, Jay N, Jones SM, Kim EH, Kloepfer K, Leonard S, Lezmi G, Lieberman J, Lomas J, Makhija M, O'Sullivan M, Parrish C, Peake J, Perrett KP, Petroni D, Pongracic JA, Quinn P, Robison RG, Sanders G, Schneider L, Sharma H, Sindher SB, Trujillo J, Turner PJ, Tuttle K, Upton J, Varshney P, Vickery BP, Vogelberg C, Wainstein B, Wang J, Wood R, Bee KJ, Campbell DE, Green TD, Rouissi R, Bahnson HT, Bois T, Sampson HA, Burks AW. Efficacy and Safety of Epicutaneous Immunotherapy in Peanut-Allergic Toddlers: Open-Label Extension to EPITOPE. J Allergy Clin Immunol Pract. 2025 May;13(5):1176-1187.e7. doi: 10.1016/j.jaip.2025.02.004. Epub 2025 Feb 14. PMID 39956162
- [Derived] Greenhawt M, Sindher SB, Wang J, O'Sullivan M, du Toit G, Kim EH, Albright D, Anvari S, Arends N, Arkwright PD, Begin P, Blumchen K, Bourrier T, Brown-Whitehorn T, Cassell H, Chan ES, Ciaccio CE, Deschildre A, Divaret-Chauveau A, Dorris SL, Dorsey MJ, Eiwegger T, Erlewyn-Lajeunesse M, Fleischer DM, Ford LS, Garcia-Lloret M, Giovannini-Chami L, Hourihane JO, Jay N, Jones SM, Kerns LA, Kloepfer KM, Leonard S, Lezmi G, Lieberman JA, Lomas J, Makhija M, Parrish C, Peake J, Perrett KP, Petroni D, Pfutzner W, Pongracic JA, Quinn P, Robison RG, Sanders G, Schneider L, Sharma HP, Trujillo J, Turner PJ, Tuttle K, Upton JE, Varshney P, Vickery BP, Vogelberg C, Wainstein B, Wood RA, Bee KJ, Campbell DE, Green TD, Rouissi R, Peillon A, Bahnson HT, Bois T, Sampson HA, Burks AW. Phase 3 Trial of Epicutaneous Immunotherapy in Toddlers with Peanut Allergy. N Engl J Med. 2023 May 11;388(19):1755-1766. doi: 10.1056/NEJMoa2212895. PMID 37163622